CLINICAL TRIAL: NCT04731038
Title: Combination of Paclitaxel, Cisplatin\Carboplatin With Toripalimab and Anlotinib for First Line Treatment of Advanced Cervical Cancer
Brief Title: Combination Therapy for First Line Treatment of Advanced Cervical Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Jun Zhang, Chair of Department of Oncology, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COMSTRAIN-CESC
Record Dates: First submitted 2021-01-27; First posted 2021-01-29 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Advanced Cervical Cancer
MeSH Terms: interventions — anlotinib; toripalimab; Paclitaxel; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Anlotinib 12mg qd. po. d1-d14 q3w Toripalimab 240mg ivgtt. d1 q3w Paclitaxel 135mg/m2 ivgtt. d1 q3w Cisplatin 50mg/m2 ivgtt. d1 q3w Carboplatin AUC=5 ivgtt. d1 q3w
  Interventions: Drug: Anlotinib, Toripalimab, Paclitaxel, Cisplatin/ Carboplatin

INTERVENTIONS:
Drug: Anlotinib, Toripalimab, Paclitaxel, Cisplatin/ Carboplatin — This is a single-arm study with all patients receiving these four drugs.

SUMMARY:
This is a single center phase 1 trail to observe safety and efficacy of Paclitaxel plus Cisplatin\Carboplatin, PD-L1 antibody Toripalimab and Anlotinib as first-line regimen to treat the patient with metastatic 、persistent or recurrent disease after radical surgery、radical platinum-based concurrent chemoradiotherapy or both (Stage IA-IVA).

DETAILED DESCRIPTION:
Advanced cervical cancer patients with metastatic, persistent or recurrent disease after radical surgery、radical platinum-based concurrent chemoradiotherapy or both will be treated by Paclitaxel plus Cisplatin\Carboplatin, PD-L1 antibody Toripalimab and Anlotinib.

ELIGIBILITY:
Inclusion Criteria:

1. female patients aged≥18 years.
2. Histologically confirmed cervical squamous cell carcinoma or adenocarcinoma, without uncontrolled pleural effusion or ascites.
3. Patients with advanced or metastatic disease who have disease progression after radical surgery、radical platinum-based concurrent chemoradiotherapy or both （Stage IA-IVA）, with measurable lesions.
4. ECOG performance status 0 or 2, expected lifetime≥3 months.
5. Adequate organ function: Absolute neutrophil count (ANC) ≥1.5x109/L, White blood count ≥3.5x109/L, Platelets ≥100x109/L, Hemoglobin (Hb) ≥100g/L, ALT/AST ≤2.5x ULN (for patient with liver metastasis ALT/AST ≤5x ULN), Serum bilirubin ≤1.5x ULN, Serum creatinine ≤1.5x ULN.
6. HBV infected patients (inactive/asymptomatic carrier, chronic or active) with HBV DNA<500IU/ml (or 2500 copies/ml).
7. Pregnancy test of female patients with fertile activity should be negative within 7 days before enrollment. Patients should keep contraception during treatment.
8. Willingness and ability to comply with the protocol for the duration of the study including scheduled visits, examinations, investigations and treatment plans with informed consent form.

Exclusion Criteria:

1. Pregnancy or children bearing potential.
2. brain or meningeal metastasis.
3. With second primary malignant diseases.
4. With uncontrolled auto-immune diseases, interstitial pneumonia, ulcerative colitis, or patients who should receive long-term glucocorticoid treatment (>10mg/d prednisone).
5. With uncontrollable complications
6. Inadequate organ function
7. Conditions which impact on pill taking (dysphagia, chronic diarrhea, bowel obstruction).
8. known hypersensitivity reaction to any of the study drugs or components.
9. Other unsuitable conditions determined by investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Safety: adverse events as assessed by CTCAE v5.0 | 36 months

SECONDARY OUTCOMES:
Progression free survival | 36 months
Overall survival | 36 months
Objective response rate | 36 months
Disease control rate | 36 months
Duration of response | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, MD & Ph. D, Principal Investigator — Ruijin Hospital
Locations (1):
- Department of Oncology, Ruijin Hospital, Shanghai, China